CLINICAL TRIAL: NCT01002092
Title: A Randomized, Controlled Multicenter Trial of Endostar Combined With Chemotherapy for Treatment of Osteosarcoma
Brief Title: A Study of Endostar Combined With Chemotherapy for Treatment of Osteosarcoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Shandong Simcere-Medgenn Bio-pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SIM-65
Record Dates: First submitted 2009-10-25; First posted 2009-10-27 (Estimated); Last update posted 2014-09-03 (Estimated); Status verified 2014-08

CONDITIONS: Osteosarcoma
Keywords: Osteosarcoma; Endostar; Chemotherapy
MeSH Terms: conditions — Osteosarcoma | interventions — Drug Therapy; endostar protein

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Chemotherapy (Active Comparator)
  Interventions: Drug: Chemotherapy
- Endostar plus Chemotherapy (Experimental)
  Interventions: Drug: Chemotherapy; Drug: Endostar

INTERVENTIONS:
Drug: Chemotherapy — Week 1 day 1 MTX 8 g/m2; Week 3 day 1-2 CDP 100-120 mg/m2 day 1 ADM/THP 60 mg/m2; Week 5 day 1-6 IFO 2 g/day; Week 7 rest; Week 8 surgery; Two weeks after the surgery repeat the chemotherapy cycle 3 times (6 weeks per cycle).
Drug: Endostar — In each cycle, Week 1-2 day 1-14 endostar 7.5 mg/m2/day; Week 5-6 day 1-14 endostar 7.5 mg/m2/day
  Arms: Endostar plus Chemotherapy

SUMMARY:
Purpose: This study will assess the safety and efficacy of Endostar combined with chemotherapy in osteosarcoma patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically confirmed osteosarcoma, who have no evidence of metastasis
* At least one measurable lesion
* Life expectancy > 3 months
* ECOG performance status 0-2
* Adequate hematologic, cardiac, renal, and hepatic function
* Patients with prior chemotherapy should have at least 4 weeks clearance period before entering this study

Exclusion Criteria:

* Evidence of metastasis
* Serious infection
* Evidence of bleeding diathesis
* Significant cardiovascular disease
* Pregnant or lactating woman
* Allergic to E.coli preparation

Ages: 12 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 160 (Estimated)
Dates: Start 2009-02; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival | 5 years

SECONDARY OUTCOMES:
Limb Salvage Rate | end of the first cycle
Overall Survival | 5 years
Clinical Response Rate | end of the first cycle
Clinical Benefit Response | end of the first cycle
Quality of Life | after 4 cycles

CONTACTS AND LOCATIONS:
Overall Officials: Sujia Wu, Dr., Principal Investigator — Nanjing PLA General Hospital; Xin Shi, Dr., Principal Investigator — Nanjing PLA General Hospital
Locations (4):
- China (4):
  - Nanjing General Hospital of Nanjing Military Command, Nanjing, Jiangsu
  - General Hospital of Jinan Military Command, Jinan, Shandong
  - Xijing Hospital, Xi’an, Shanxi
  - The Military General Hospital of Beijing PLA, Beijing